CLINICAL TRIAL: NCT01237665
Title: A Phase II Trial of Neoadjuvant IXO Regimen (Irinotecan, Capecitabine [Xeloda], Oxaliplatin) Followed by Combined Modality Capecitabine and Radiation for Locally Resectable Advanced Rectal Cancer
Brief Title: IXO (Irinotecan, Xeloda, Oxaliplatin) in Rectal Cancer
Acronym: IXOr
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Ottawa Regional Cancer Foundation (Unknown); Sanofi (Industry); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OTT 09-02
Record Dates: First submitted 2010-08-25; First posted 2010-11-09 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Rectal Cancer
Keywords: locally resectable advanced adenocarcinoma of the rectum
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IXO regimen (Experimental): single-group
  Interventions: Drug: IXO regimen

INTERVENTIONS:
Drug: IXO regimen — IXO regimen is administered as following: irinotecan 160 mg/m2 i.v. (over 60-90 minutes) with oxaliplatin 100 mg/m2 i.v. (over 120 minutes) on day 1, followed by capecitabine 950 mg/m2 PO, b.i.d. on days 2-15, every 3 weeks.
  Each cycle of IXO lasts 21 days, with the subsequent cycle to start on day 22.

SUMMARY:
This is a prospective open label single-arm, single-institution phase II clinical trial to test the efficacy of neoadjuvant treatment with IXO (Irinotecan, Capecitabine [Xeloda], Oxaliplatin) followed by chemoradiotherapy and resection in patients with resectable non-metastatic primary rectal cancer of stage cT3-T4 N0-N2.

ELIGIBILITY:
Inclusion Criteria:

General

* Pathologically confirmed rectal adenocarcinoma
* T3 or T4 or N1 (node ≥1 cm on short axis) adenocarcinoma of the rectum.
* ECOG performance status equal or less than 1
* Male and female patients, aged ≥ 18 years and ≤ 80 years
* Written informed consent
* Adequate haematological, liver, renal function

Resectability

* Patients categorized as having resectable locally advanced cancer
* Favorable general condition

Exclusion Criteria:

Resectability

* Diagnosis of metastatic disease
* Clear indication of involvement of pelvic wall(s), on imaging.
* Peritoneal carcinomatosis, portal vein occlusion, ascites, non-regional lymph nodes
* Histology other than adenocarcinoma
* Obstructed rectal carcinoma without defunctionalizing colostomy

Prior treatment

* Previously undergone treatment for this disease
* Prior chemotherapy for colorectal cancer
* Prior chemotherapy for other malignancies in past 12 months
* Prior radiotherapy other than skin cancer
* Concomitant use of St John's Wort
* Treatment with any other investigational agent
* Current use of full-dose of warfarin for therapeutic

Other conditions

* Confirmed or suspected brain metastases
* History or evidence of CNS disease
* Past or current history of other malignancies
* Clinically significant cardiovascular disease
* Evidence of bleeding diathesis or coagulopathy
* Known hypersensitivity to any of the study drugs
* Serious, non-healing wound, ulcer or bone fracture
* Major surgical procedure or significant traumatic injury within 28 days prior to treatment
* Disease or condition that contraindicates the use of an investigational drug
* Life expectancy less than 5 years
* Inability or unwillingness to comply with the protocol
* Neuropathy ≥ Gr.2
* History of ulcerative colitis or Crohn's disease
* Pelvic abscess or perforated pelvic carcinoma

Pregnancy / Contraception

* Pregnancy or lactation
* Positive serum pregnancy test within 7 days of starting study treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) | 26 weeks
  To test the efficacy of neoadjuvant treatment with IXO followed by chemoradiotherapy and surgical resection, evaluated as histological therapy-induced tumour regression, assessed by the rate of pathological complete response (pCR) at the primary tumor site (pT0)

SECONDARY OUTCOMES:
Objective Response | 12 weeks and 18 weeks
  Objective Response by MRI - post IXO and post RCT
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | every 3 weeks during neoadjuvant chemotherapy; before CRT; 3rd week of CRT; 2 days, 3 weeks and 6 weeks post CRT; pre-op; 2 days and 4 weeks post-op
  Toxicity according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) v.3.0 and drug safety
Recurrence | q6 months
  Rates of local and distant disease recurrence
RFS, PFS, TTR | q6 months
  Recurrence free survival (RFS), progression free survival (PFS), time to recurrence (TTR)
Quality of life | enrolment, 12 weeks, 18 weeks, 26 weeks
  Quality of life (QoL) as assessed by the EORTC QLQ-C30 scale
Surgical morbidity and mortality | 26 weeks
  post-operative
Rate of post-operative sphincter preservation | 26 weeks
  post-operative
OS | q6 months first 2 years and annually thereafter
  overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Derek Jonker, MD, Principal Investigator — The Ottawa Hospital Cancer Centre
Locations (1):
- The Ottawa Hospital Cancer Centre, Ottawa, Ontario, Canada